CLINICAL TRIAL: NCT05729373
Title: A Phase 2/3, Randomized, Double-blind, Parallel Group, Placebo-controlled, Flexible-dose, Multicenter Study to Evaluate the Efficacy and Safety of SEP-363856 in the Treatment of Adults With Generalized Anxiety Disorder
Brief Title: A Clinical Study That Will Measure How Well SEP-363856 Works and How Safe it is in Adults With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP361-226; 2022-502077-42-00 (Other: EMA); jRCT2031230152 (Registry Identifier: Japan Registry for Clinical Trials (jRCT))
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — SEP-363856

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Parallel group, Placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SEP-363856 (Experimental): dosed once daily tablet
  Interventions: Drug: SEP-363856
- Placebo (Placebo Comparator): dosed once daily tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SEP-363856 — once daily tablet
  Arms: SEP-363856
Drug: Placebo — once daily tablet
  Arms: Placebo

SUMMARY:
A clinical study that will meaure how well SEP-363856 works and how safe it is in adults with Generalized Anixety Disorder. This study will be accepting both male and female subjects between the ages of 18 years and 65 years old. The study will be held in Approximately 50 global study centers and approximately 15 additional centers for a separate Japan population. Participation in the study can be up to approximately 12 weeks.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel-group, flexible dose, outpatient study evaluating the efficacy and safety of SEP-363856 flexibly dosed (50 - 75 mg/day) versus placebo over an 8-week Treatment Period in subjects with GAD. This study is projected to randomize approximately 434 subjects to 2 treatment groups (SEP-363856 [50 - 75 mg/day] or placebo) in a 1:1 ratio.

Approximately 30 additional subjects (N = 15 per treatment group) are projected to enroll in the Japan Cohort. Treatment assignment will be stratified by country. Study drug will be taken at approximately the same time each evening at bedtime .

ELIGIBILITY:
Inclusion Criteria: (list is not all inclusive)

* Male or female subject between 18 to 65 years of age.
* Subject meets DSM-5 criteria for a diagnosis of Generalized Anxiety Disorder.
* Subject must be willing and able to comply with the study procedures and visit schedule and must be able to understand and follow verbal and written instructions.

Exclusion Criteria: (list is not all inclusive)

* Subject has DSM-5-based diagnosis of any disorder other than Generalized Anxiety Disorder that was the primary focus of treatment within 12 months before Screening.
* Subjects who report an inadequate response to more than 3 antidepressant treatments
* Subject is at significant risk of harming self or others based on Investigator's judgment.
* Subject has any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study.
* Female subject who is pregnant, lactating, or plans to get pregnant during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Hamilton Anxiety Rating Scale (HAM-A) total score at Endpoint | Week 8
  The HAM-A scale consists of 14 items, each defined by a series of symptoms. Each item is rated on a 5-point (0-4) scale, with higher scores indicating greater severity.

SECONDARY OUTCOMES:
Change from Baseline in Clinical Global Impression-Severity (CGI-S) score at Endpoint | Week 8
  The CGI-S is a clinician-rated assessment of the subject's current illness state on a 7-point scale, where a higher score is associated with greater illness severity.

CONTACTS AND LOCATIONS:
Locations (83):
- United States (38):
  - University of Alabama at Birmingham, Huntsville, Alabama
  - IMA Clinical Research Phoenix, Phoenix, Arizona
  - ProScience Research Group, Culver City, California
  - Excell Research, Inc., Oceanside, California
  - Anderson Clinical Research, Redlands, California
  - California Neuroscience Research, LLC, Sherman, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Viking Pharmaceutical Trials Inc. dba Viking Clinical Research, Temecula, California
  - CenExel Collaborative Neuroscience Research, Torrance, California
  - Pacific Clinical Research Management Group, Upland, California
  - CNS Healthcare, Jacksonville, Florida
  - Combined Research Orlando, Orlando, Florida
  - K2 Medical Research, LLC, Tampa, Florida
  - CenExel iResearch Atlanta, Atlanta, Georgia
  - Advanced Discovery Research LLC, Atlanta, Georgia
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - CenExel iResearch Savannah, Savannah, Georgia
  - Uptown Research Institute, LLC, Chicago, Illinois
  - American Medical Research, Inc., Warrenville, Illinois
  - Copley Clinical, Boston, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Midwest Research Group, Saint Charles, Missouri
  - Center for Emotional Fitness Site, Cherry Hill, New Jersey
  - CenExel Hassman Research Institute, Marlton, New Jersey
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Bioscience Research, LLC, Mount Kisco, New York
  - Berman Clinical, New York, New York
  - Manhattan Behavioral Medicine, New York, New York
  - The Medical Research Network, L.L.C, New York, New York
  - Neuro-Behavioral Clinical Research, Inc., North Canton, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, LLP, Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research, LLC, Allentown, Pennsylvania
  - Psychiatry and Psychotherapy Partners Austin, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Cedar Clinical Research, Inc., Draper, Utah
- Bulgaria (9):
  - Medical Center Mentalcare OOD, Sofia, Plovdiv
  - Medical Center Medconsult Pleven OOD, Pleven
  - MHC - Sofia, EOOD, Sofia
  - Medical Center "Sv.Naum", Sofia
  - DCC "Sv. Vrach and Sv. Sv. Kuzma and Damyan", OOD, Sofia
  - Medical Center Hera EOOD, Sofia
  - Medical Center Intermedica, OOD, Sofia
  - DCC "Mladost M" - Varna, OOD Site #156, Varna
  - DCC "Mladost M" - Varna, OOD Site #157, Varna
- Estonia (2):
  - Marienthali Kliinik, Tallinn
  - Tartu University Hospital, Tartu
- Finland (5):
  - Savon Psykiatripalvelu Oy, Kuopio, Northern Savonia
  - Aava Laakarikeskus - Aava Kamppi, Helsinki
  - Mederon Oy, Helsinki
  - Oulu Mentalcare Oy, Oulu
  - Satakunnan Psykiatripalvelu, Tampere
- Japan (14):
  - Uematsu Mental Clinic, Chikugo-shi, Fukuoka
  - Hiro Mental Clinic, Fukuoka, Fukuoka
  - Shinseikai Kaku Mental Clinic, Fukuoka, Fukuoka
  - Mental Clinic Sakurazaka, Fukuoka, Fukuoka
  - Kokura Mental Clinic, Kitakyushu-shi, Fukuoka
  - Hirota Clinic, Kurume-shi, Fukuoka
  - Hayakawa Clinic, Kure-shi, Hiroshima
  - Higashi-Sapporo Mental Clinic, Sapporo, Hokkaido
  - Shimode Mental Clinic, Sapporo, Hokkaido
  - Akari Clinic, Naha, Okinawa
  - Barclay Imuro Mental Clinic, Urasoe-shi, Okinawa
  - Senzoku Psychosomatic Medicine Clinic, Meguro-ku, Tokyo-To
  - Sangenjaya Nakamura Mental Clinic, Setagaya-ku, Tokyo-To
  - Sangenjaya Neurology- Psychosomatic Clinic, Setagaya-ku, Tokyo-To
- Slovakia (5):
  - MENTUM, s.r.o., Bratislava
  - Epamed sro, Košice
  - PsychoLine s.r.o., Rimavská Sobota
  - Crystal Comfort s.r.o., Vranov nad Topľou
  - BONA MEDIC, s.r.o., Zlaté Moravce
- Spain (6):
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Valle del Nalon, Langreo, Principality of Asturias
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Institucion Hospitalaria Hestia Palau, Barcelona
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital de Antequera, Málaga
- Sweden (4):
  - Sahlgrenska Universitetssjukhuset - Östra sjukhuset, Gothenburg
  - ProbarE- Lund, Lund
  - PharmaSite AB Malmö, Malmo
  - ProbarE- Stockholm, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com